CLINICAL TRIAL: NCT04541836
Title: Image Characteristic and Longitudinal Follow up of 18F-PMPBB3 (APN-1607) PET for Progressive Supranuclear Palsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201901999A0
Record Dates: First submitted 2020-08-31; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Progressive Supranuclear Palsy
Keywords: tauopathy; Progressive Supranuclear Palsy; F-18 APN1607 PET; F-18 PMPBB3 PET
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Tauopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy control: healthy volunteer with no clinically relevant finding on physical examination at screening visit will receive one baseline 18F-PMPBB3 tau PET scan, and another follow up scan 1.5yr later.
  Interventions: Diagnostic Test: 18F-PMPBB3
- PSP: Patients fulfill the criteria of NINDS-SPSP clinical criteria for the diagnosis of PSP "as possible" or "probably" PSP will receive one baseline 18F-PMPBB3 tau PET scan, and another follow up scan 1.5yr later.
  Interventions: Diagnostic Test: 18F-PMPBB3

INTERVENTIONS:
Diagnostic Test: 18F-PMPBB3 — single intravenous injection 5mCi 18F-PMPBB3 per scan
  Other Names: 18F-APN-1607; 18F-MNI-958; 18F-APN-0000455

SUMMARY:
The study will enroll 20 PSP and 8 normal subjects with complete neurological examination, 18F-PMPBB3 (APN-1607) PET and MRI assessment. To explore: (1) whether 18F-PMPBB3 (APN-1607) can detect the 4R tau protein in the brain of PSP patients; (2) whether 18F-PMPBB3 (APN-1607) can distinguish the clinical characteristics of PSP; (3) Whether the distribution of tau deposition is related to disease severity, progression, and prognosis.

DETAILED DESCRIPTION:
Progressive supranuclear palsy (PSP), also known as Steele-Richardson-Olszewski syndrome, has a similar incidence in men and women. The pathophysiology of PSP is remaining unclear, but it is known to be related to the abnormal accumulation of 4R tau protein in the brain. Recently, new generation of novel radiotracer 18F-PMPBB3 (APN-1607), which can be labeled with 4R PHF-tau without significant off-target binding, has been successfully developed. The study will enroll 20 PSP and 8 normal subjects with complete neurological examination, 18F-PMPBB3 (APN-1607) PET and MRI assessment. To explore: (1) whether 18F-PMPBB3 (APN-1607) can detect the 4R tau protein in the brain of PSP patients; (2) whether 18F-PMPBB3 (APN-1607) can distinguish the clinical characteristics of PSP; (3) Whether the distribution of tau deposition is related to disease severity, progression, and prognosis. The research results will help to understand the potential of 18F-PMPBB3 (APN-1607) as a biomarker for diagnosis and therapeutic assessment tool for progressive nuclear paralysis as well as other tau proteinopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Patients fulfill the criteria of NINDS-SPSP clinical criteria for the diagnosis of PSP "as possible" or "probably" PSP, and healthy volunteer with no clinically relevant finding on physical examination at screening visit.
3. Age range 20-90 years

Exclusion Criteria:

1. Implantation of metal devices including cardiac pacemaker, intravascular metal devices.
2. Major systemic diseases including coronary arterial disease, heart failure, uremia, hepatic failure, prominent strokes, acute myocardial infarction, poorly controlled diabetes, previous head injury, intracranial operation, hypoxia, sepsis or severe infectious diseases
3. Major psychiatric disorders, drug or alcohol abuse and major depression
4. Pregnant women or breast- feeding women

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PSP patient will be enrolled from primary care clinic or hospital, control (healthy subjects) will be enrolled from community.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Tau Distribution Among Progressive Supranuclear Palsy (PSP), and Normal Subjects | 5 days
  Tau Distribution Among Progressive Supranuclear Palsy (PSP), and Normal Subjects Measured by Standardized Uptake Value Ratio (SUVR) as Assessed by 18F-PM-PBB3 tau PET Scan

SECONDARY OUTCOMES:
To assess disease severity in PSP | 5 days
  To assess disease severity in PSP subjects by SUVR as Assessed by 18F-PM-PBB3 tau PET Scan
To assess disease progression in PSP | 1.5 year
  To assess disease progression in PSP subjects by SUVR as Assessed by 18F-PM-PBB3 tau PET Scan
Blood pressure | 3 hours
  Systolic and diastolic pressure of subjects will be measured right before injection and after scanning.
Pulse | 3 hours
  Pulse will be measured right before injection and after scanning.
Respiration frequency | 3 hours
  Respiration frequency will be measured right before injection and after scanning.
Adverse events collection | 5 days
  Adverse events within 5 days after the injection and scanning of subjects will be followed and assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital,Linkou, Taoyuan, Guishan Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No
no plan